CLINICAL TRIAL: NCT06711250
Title: Repeated Injection of I PRF and Autogenous Bone Graft for Alveolar Ridge Augmentation :randomized Controlled Clinical Trial
Brief Title: Repeated Injection of I PRF and Autogenous Bone Graft for Alveolar Ridge Augmentation
Acronym: I-PRF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: alveolar ridge augmenation
Record Dates: First submitted 2024-11-22; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Alveolar Bone Loss; Alveolar Ridge Abnormality
Keywords: A lveolar ridge defect , Khoury technique Guided bone regeneration, i PRF, CBCT analysis
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control (Active Comparator): bone grafting
  Interventions: Procedure: khoury technique
- study (Active Comparator): bone grafting & i PRF
  Interventions: Procedure: khoury technique with i-PRF injections

INTERVENTIONS:
Procedure: khoury technique — autogenous bone augmentation
  Arms: control
Procedure: khoury technique with i-PRF injections — autogenous bone augmentation with repeated i-PRF injections
  Arms: study

SUMMARY:
The current st udy's objective was to validate the repeated effect of i PRF with autogenous bone on the of gingival thickness , width a n d volumetric bone changes durig maxillary alveolar augmentation using cone beam computer tomography (CBCT). Patients and methods:

DETAILED DESCRIPTION:
The study was a randomized clinical study in which participants needed to augment defective ridge were selected from the Outpatient Clinic, Department of Oral Medicine, Periodontology and Diagnosis , Faculty of Dental Medicine for Girls, Al Azhar University. The Research Ethics Committee, Faculty of Dental Medicine for Girls, Al Azhar University (REC code (P. PD 24 19 ) certified this study and a signed informed consent form with approval was obtained from each. Each patient who was enrolled in the study had a complete medical record and a proper clinical examination. These patients had to have a horizontal or vertical alveolar ridge deficiency and have enough bone in the mandibular donor site (external oblique ridge).

However, patients showing any signs of active periodontal disease, on long term corticosteroid therapy, persons taking bone metabolism drugs as well as individuals suffering from any systemic illness that may impact bone repair were excluded from the study.

Patients were assigned to one of two 2 groups, group I or group II. Group I, consisted of patients grafted with autogenous bone graft alone. I n Group II, patients were grafted using autogenous bone combined with repeated injection of i PRF Assessment of the alveolar ridge dimension and the bone block to be harvested preoperatively using CBCT. T he measurements of the alveolar ridge mesio distaly and bucco lingually in mm were determined at the recipient site . It was crucial to visualize the anatomic structures at the osteotomy site, including the alveolar canal, the mental foramina, and the teeth roots present to create ideal bone cutting planes according to the depth and extension of the graft without any injuries to the aforementioned structures.

ELIGIBILITY:
Inclusion Criteria:

* patients who have a horizontal or vertical alveolar ridge deficiency

Exclusion Criteria:

* patients showing any signs of active periodontal disease
* patients on long term corticosteroid therapy,
* patients taking bone metabolism drugs
* patients suffering from any systemic illness that may impact bone repair

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
width of the alveolar ridge | baseline, 6 months & 9 months
  CBCT will be used to assess the width of the alveolar ridge

SECONDARY OUTCOMES:
volumetric analysis of bone | at baseline, 6 and 9 months
  volumetric analysis ob bone using CBCT to assess the bone volume

CONTACTS AND LOCATIONS:
Overall Officials: Zainab H Abdel Rahman, Phd, Principal Investigator
Locations (1):
- Faculty of Dentistry , Al Azhar Univeristy For Girls, Cairo, Heliopolis - Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No